CLINICAL TRIAL: NCT05155059
Title: Phase II Trial of Non-Invasive Intermittent Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex in Functional Movement Disorders
Brief Title: Non-invasive Intermittent Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex in Functional Movement Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10000642; 000642-N
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05-30

CONDITIONS: Functional Movement Disorder
Keywords: Functional Movement Disorders; Transcranial Magnetic Stimulation (TMS); iTBS; Repetitive Transcranial Magnetic Stimulation; Neuroimaging; Conversion Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Sham TMS stimulation using a sham coil
  Interventions: Other: Sham Comparator
- Treatment (Experimental): Active TMS stimulation using an active TMS coil
  Interventions: Device: MagStim

INTERVENTIONS:
Device: MagStim — Bursts of three at 50Hz with an inter burst interval of 200 ms will be given for 190 seconds and this session will be repeated 3 times with 20 minutes between each session in one day. The set of 3 sessions will be repeated 5 times in 5 consecutive days.
  Arms: Treatment
Other: Sham Comparator — Sham TMS stimulation using a sham coil
  Arms: Control

SUMMARY:
Background:

Functional movement disorders (FMD) involve involuntary movements that are not due to a recognized neurological or medical cause. FMD can cause major disability. Researchers want to learn more to create better treatments for FMD.

Objective:

To test whether non-invasive brain stimulation using transcranial magnetic stimulation (TMS) improves FMD symptoms.

Eligibility:

People between the ages of 18 and 80 who have been diagnosed with FMD by a neurologist.

Design:

Participants will be randomly assigned to one of two groups. One group is an active brain stimulation group and the other is a sham brain stimulation group.

Participants will have a baseline visit. This will include:

Neurological exam

Questionnaires

Urine test

Brain MRI: Participants will lie in a machine that takes pictures of the body. They will be asked to respond to images on a screen while in the scanner.

Within 2 weeks of the baseline visit, participants will begin 5 daily sessions of TMS. The active group will have stimulation delivered to the brain via a coil. In the sham group, a dummy coil will be used that will not deliver stimulation. A total of three 3-minute cycles will be done in one visit. There will be 20-minute breaks between the cycles.

Participants will have visits 1 month, 2 months, and 6 months after their last day of TMS. Their FMD symptoms will be evaluated. They will complete health questionnaires. These visits can be in person or virtual.

DETAILED DESCRIPTION:
Study Description:

The purpose of this protocol is to investigate efficacy of intermittent theta burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC) in patients with functional movement disorders (FMD). Participants will be randomly assigned to receive either active iTBS or sham stimulation of the left DLPFC for 5 consecutive daily sessions.

Objectives:

Primary Objective: To investigate efficacy of iTBS of the left DLPFC on motor symptoms in patients with FMD

Secondary Objectives: To investigate efficacy of iTBS of the left DLPFC on mood symptoms and its effect on fronto-amygdala circuit on functional neuroimaging

Endpoints:

Primary Endpoint: Relative change in Functional Movement Disorder Rating Scale (S-FMDRS) from the baseline to 1 month after iTBS vs sham: 100 *( S-FMDRS at one-month - S-FMDRS at baseline)/ S-FMDRS at baseline

Secondary Endpoints:

* S-FMDRS immediately after, 2 months and 6 months after the treatment
* HADS at 1 month, 2 months and 6 months after the treatment
* DLPFC-amygdala functional connectivity
* Amygdala BOLD response to emotional stimuli

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-80
* Diagnosis of functional movement disorder made by a neurologist
* Agreement to adhere to Lifestyle Considerations throughout study duration
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Current psychosis or active suicidal ideation
* History of epilepsy with the exception of febrile seizure
* Patients with psychogenic non-epileptic seizure without comcomitant functional movement disorder
* Any significant neurological disorders other than FMD including but not limited to multiple sclerosis, stroke, Parkinson s disease, space occupying brain lesion
* Alcohol or substance use disorder
* Patients who are on Buproprion (Wellbutrin)
* Patients with moderate to severe cardiac disease
* Any psychiatric, medical or social condition due to which, in the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
S-FMDRS | 1 month after iTBS
  Short version of Functional Movement Disorder Rating Scale

SECONDARY OUTCOMES:
S-FMDRS | 2 and 6 months after iTBS
  Short version of Functional Movement Disorder Rating Scale
SF-36 | 1, 2 and 6 months after iTBS
  Health related quality of life
CGI | 1, 2 and 6 months after iTBS
  Clinical Global impression - scale of 1-7 to measure clinical improvement from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD during the trial can be shared after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 2 years after the publication
Access Criteria: IPD can be shared with researchers who provide methodologically sound proposal for meta-analysis or any other scientific analysis. Requests should be directed to the study PI who will review requests. Only de-identified data will be shared for scientific purposes.

REFERENCES:
- [Background] Spagnolo PA, Parker J, Horovitz S, Hallett M. Corticolimbic Modulation via Intermittent Theta Burst Stimulation as a Novel Treatment for Functional Movement Disorder: A Proof-of-Concept Study. Brain Sci. 2021 Jun 15;11(6):791. doi: 10.3390/brainsci11060791. PMID 34203993
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000642-N.html